CLINICAL TRIAL: NCT05787782
Title: Validation of the Masimo INVSENSOR00063 in Febrile and Afebrile Subejcts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KOEI0004
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2023-06

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Masimo INVSENSOR00063 (Experimental): All subjects are enrolled into this arm and will have temperature measurements obtained.
  Interventions: Device: Masimo INVSENSOR00063

INTERVENTIONS:
Device: Masimo INVSENSOR00063 — Masimo INVSENSOR00063 will be used to measure temperature

SUMMARY:
This is a prospective, non-randomized data collection study to evaluate the performance of the Masimo INVSENSOR00063 in obtaining temperature measurements.

DETAILED DESCRIPTION:
Individual sites are only representative of a subset of the overall population, per ISO 80601-2-56:2017(Medical electrical equipment - Part 2-56: Particular requirements for basic safety and essential performance of clinical thermometers for body temperature measurement), and therefore clinical bias and limits of agreement should not be evaluated for the subsets. Publication of results should include repeatability from individual sites and the combined clinical bias and limits of agreement (NCT05787782, NCT05674344 and NCT05779397).

ELIGIBILITY:
Inclusion Criteria:

* Participant age ≥ 1 year
* Afebrile or febrile at time of enrollment: For febrile subjects, ≥ 99.5 F/ 37.5 C for sublingual temperature reference; ≥ 100.4 F/ 38 C for temporal artery temperature reference.
* English-or Spanish-speaking patient or parent/Legal Guardian

Exclusion Criteria:

* Participants deemed not suitable for the study at the discretion of the investigator

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ascada Research, Fullerton, California, United States

REFERENCES:
- See also: Calibration and Validation of the Masimo Rad-G with Temperature device in Febrile Patients — https://clinicaltrials.gov/ct2/show/NCT05674344?term=choc0008&draw=2&rank=1
- See also: Clinical Performance of Masimo Rad-GT — https://clinicaltrials.gov/ct2/show/NCT05779397?term=CIP-1064&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Masimo INVSENSOR00063
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Masimo INVSENSOR00063
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31
  Between 18 and 65 years | 28
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 9
  White | 38
  More than one race | 5
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Temperature Measurements Using Masimo INVSENSOR00063
Description: Masimo INVSENSOR00063 temperature measurements will be compared to reference temperature measurements. Accuracy of Masimo INVSENSOR00063 will be measured using clinical bias, limits of agreement and repeatability.
Time Frame: About 15-30 minutes
Population: Data for 1 subject was excluded as they did not complete one round of measurements.
  Data for 1 subject was excluded as the data suggested existence of external conditions that interefere with RCT (reference clinical thermometer) or Masimo INVSENSOR00063 measurements.
Measure: Number; unit: Degrees Celsius
Arm/Group | Masimo INVSENSOR00063
Number analyzed (Participants) | 58
Degrees Celsius
  Clinical Bias | -0.24
  Limits of Agreement | 0.85
  Repeatability | 0.05

ADVERSE EVENTS:
Time Frame: 15-30 minutes during data collection
Arm/Group | Masimo INVSENSOR00063
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT05787782/Prot_SAP_000.pdf